CLINICAL TRIAL: NCT00855699
Title: Alcohol Detoxification in Primary Care Treatment (ADEPT) - a Feasibility Study of Conducting a Randomised Trial in Primary Care Comparing Two Pharmacological Regimens.
Brief Title: Alcohol Detoxification in Primary Care Treatment (ADEPT)
Acronym: ADEPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bristol (Other)
Responsible Party: Dr Anne Lingford-Hughes, University of Bristol
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RED 740; RfPB: PB-PG-0407-13296; EUDRACT: 2008-004820-22
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Alcoholism
Keywords: Alcohol detoxification
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Acamprosate — Acamprosate 333mg tablets, two tablets three times a day for duration of alcohol detox.
  Other Names: Campral

SUMMARY:
Once someone becomes dependent on alcohol (alcoholic), the risks of complications from alcohol withdrawal when they stop drinking grow. These can include a life-threatening fit or delirium tremens (see things, become frightened). To prevent such complications, people take medication such as benzodiazepines (e.g., valium or librium) in reducing doses for about a week; this is called detoxification or 'detox.' In the UK effective alcohol treatment exists but little is known about what is the best detox medication. Alternative drugs to benzodiazepines appear to protect the brain from the toxicity of alcohol withdrawal and to reduce the likelihood of drinking again. This study will examine the feasibility of comparing medication regimens for alcohol detox for the first time in primary care. It will include a standard detox regimen (librium over 8 days) alone and together with a drug, acamprosate, that has been shown to reduce toxicity of alcohol withdrawal in preclinical models and is used after detox to help people remain sober. It will focus on the practicalities of doing such a study as well as assessing how people feel (withdrawal symptoms) and do (drinking during first month).

DETAILED DESCRIPTION:
Aims and objectives:

To provide a framework for investigating the hypothesis that for those patients undergoing alcohol detox in primary care adding acamprosate to a reducing regimen of a benzodiazepine (chlordiazepoxide) provides better symptom control during detox compared with benzodiazepine alone. In addition we will assess improvement in sleep, drinking outcomes, completion rates and cognitive performance.

Specific primary aim:

This feasibility study aims to inform a full application for an RCT to compare the effectiveness and cost-effectiveness of acamprosate as an adjunctive treatment for benzodiazepines for alcohol detox in primary care.

Key objectives are to:

1. determine the optimal method of recruiting patients in primary care and estimate likely recruitment rate
2. investigate feasibility of completion of and variation in our proposed primary outcome measure in the community - Clinical Institute of Withdrawal Scale-Alcohol (symptoms during detox), and secondary outcome measures - drinking during first month (via diary to derive % days abstinent), completion of detox, sleep and cognitive performance.
3. investigate patient and GP acceptability of this randomised trial using qualitative measures.

ELIGIBILITY:
Inclusion Criteria:

* Anyone (18-65 years old) consulting their GP for whom a community based alcohol detox requiring medication is appropriate.
* Due to acamprosate's license for maintaining abstinence, nobody under the age of 18 and over 65 will be recruited.

Exclusion Criteria:

* Unsuitable for home/community detox, e.g., with current or significant history of:

  * delirium tremens or seizures
  * current or history of high dose polydrug use
  * significant medical or psychiatric ill health
  * pregnant or breast feeding
  * Wernicke's encephalopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Reduction in alcohol withdrawal symptoms | up to 10 days

SECONDARY OUTCOMES:
alcohol drinking | within 4 weeks of end of detox

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lingford-Hughes, Principal Investigator — University of Bristol
Locations (1):
- University of Bristol, Bristol PCT., Bristol, United Kingdom